CLINICAL TRIAL: NCT06090539
Title: A Phase 1/2, Multi-Center, Open-Label, Dose-Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BMS-986458, Alone and in Combination With Anti-lymphoma Agents in Participants With Relapsed/Refractory Non-Hodgkin Lymphomas (R/R NHL)
Brief Title: A Study to Assess BMS-986458 Alone and in Combination With Anti-lymphoma Agents in Relapsed/Refractory Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA123-1000
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A1 (Experimental): Single Agent
  Interventions: Drug: BMS-986458
- Part A2 (Experimental): Combination Treatment
  Interventions: Drug: BMS-986458; Drug: Rituximab; Drug: Glofitamab/Obinutuzumab; Drug: Mosunetuzumab
- Part B1 (Experimental): Single Agent
  Interventions: Drug: BMS-986458
- Part B2 (Experimental): Combination Treatment
  Interventions: Drug: BMS-986458; Drug: Rituximab; Drug: Glofitamab/Obinutuzumab; Drug: Mosunetuzumab

INTERVENTIONS:
Drug: BMS-986458 — Specified dose on specified days.
Drug: Rituximab — Specified dose on specified days.
  Arms: Part A2; Part B2
Drug: Glofitamab/Obinutuzumab — Specified dose on specified days
  Arms: Part A2; Part B2
Drug: Mosunetuzumab — Specified dose on specified days
  Arms: Part A2; Part B2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, and preliminary biological and clinical activity of BMS-986458, a bifunctional cereblon-dependent ligand-directed degrader of B-cell lymphoma 6 (BCL6), as a single agent and in combination with anti-lymphoma agents in participants with relapsed/refractory non-Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age with R/R NHL (including DLBCL [ie, DLBCL not otherwise specified (NOS) and diffuse large B-Cell lymphoma/high-grade B-Cell lymphoma with MYC and BCL2 rearrangements], and FL):

  * For R/R DLBCL (de novo) and FL 3b: following at least 2 prior lines of therapy (eg, first-line combination chemotherapy regimen containing rituximab, anthracycline, an alkylating agent, and steroids and at least one additional treatment).
  * For R/R DLBCL (transformed lymphoma): following at least 2 prior lines of therapy which must have been administered after transformation.
  * For R/R FL (except for FL 3b): following at least 2 prior lines of therapy and meeting treatment criteria at the time of enrollment based on investigator´s assessment.
* Participant must have measurable disease (defined by at least one FDG-avid lesion for FDG-avid disease and one bi-dimensionally measurable disease on cross sectional imaging by computed tomography or magnetic resonance imaging with at least one lesion > 1.5 cm in the transverse diameter).
* Participants must accept and follow pregnancy prevention plan.

Exclusion Criteria:

* Participants must not have an Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.
* Participants with an inability to comply with listed restrictions, precautions and prohibited treatments.
* Participants must not have prior CAR-T, or radiotherapy ≤ 4 weeks, systemic anticancer treatment ≤ 5 half-lives or 4 weeks, allogeneic SCT ≤ 6 months (only applicable to BMS-986458 single agent or rituximab combination cohorts), or autologous SCT ≤ 3 months prior to study intervention initiation.
* In BMS-986458 + T-cell engager combination cohorts: Participants must not have prior alloSCT or solid organ transplantation, history of confirmed progressive multifocal leukoencephalopathy (PML); known or suspected history of hemophagocytic lymphohistiocytosis (HLH); known or suspected chronic active Epstein-Barr (EBV) infection.
* Participants must not have any condition, including significant acute or chronic medical illness, active or uncontrolled infection, or the presence of laboratory abnormalities, that places participants at unacceptable risk if participating in this study.
* Participants must not have known or suspected central nervous system involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2028-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 2 years and 1 month
Number of participants with serious adverse events (SAEs) | Up to 2 years and 1 month
Number of participants with AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | Up to Day 28
Number of participants with AEs leading to discontiunation | Up to 2 years and 1 month
Number of participants with AEs leading to death | Up to 2 years and 1 month

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 4 months
Time of maximum concentration (Tmax) | Up to 4 months
Area under the plasma concentration-time curve within a dosing interval [AUC(TAU)] | Up to 4 months
Number of participants with a complete response rate (CRR) according to the Lugano response criteria for Non-Hodgkin Lymphoma by Investigator assessment | Up to 2 years
Number of participants with an overall response rate (ORR) according to the Lugano response criteria for Non-Hodgkin Lymphoma by investigator assessment | Up to 2 years
Duration of response (DOR) | Up to 3 years
Time to response (TTR) | Up to 3 years
Progression-free survival (PFS) | Up to 3 years
Overall survival (OS) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (12):
  - Local Institution - 0067, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Local Institution - 0068, Jacksonville, Florida
  - Local Institution - 0027, Tampa, Florida
  - Local Institution - 0014, Fairway, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0066, Rochester, Minnesota
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0040, Pittsburgh, Pennsylvania
  - Local Institution - 0045, Providence, Rhode Island
  - Local Institution - 0024, Milwaukee, Wisconsin
- France (7):
  - Local Institution - 0057, Bordeaux, Aquitaine
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Gustave Roussy, Villejuif, Paris
  - Henri Mondor Hospital, Créteil, Val-de-Marne
  - CHU SAINT ELOI - Departement Hematologie Clinique, Montpellier
  - Local Institution - 0058, Paris
  - Institut Claudius Regaud, Toulouse
- Germany (5):
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Helios Klinikum Berlin-Buch, Berlin
  - Local Institution - 0070, Essen
- Netherlands (2):
  - Maastricht UMC+, Maastricht, Limburg
  - University Medical Center Groningen, Groningen
- Spain (6):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0069, Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
- Switzerland (3):
  - Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino
  - University Hospital Basel, Basel
  - Hopitaux Universitaires de Geneve (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/ disclosure-commitment.html

REFERENCES:
- [Derived] Mortensen DS, Shunatona HP, Holmberg-Douglas N, Rhodes J, Da Silva D, Gamez J, Groza M, Zhu J, Christoforou A, Johnson SA, Khambatta G, Narla RK, Nimje RY, Huang D, Dodd DS, Griffin J, Miseo G, Whitefield B, Weiss DR, Rader J, Kuzu E, Leisten J, Lai C, Shi L, Del Rosario J, Dalvie D, Rolfe M, Zapf CW, Belmont P, Alexander M, Bence N, Groocock L. Discovery of BMS-986458, a Potent and Selective B-Cell Lymphoma 6 Protein Ligand-Directed Degrader, for the Treatment of B-Cell Non-Hodgkin Lymphoma. J Med Chem. 2026 Feb 11. doi: 10.1021/acs.jmedchem.5c03123. Online ahead of print. PMID 41670385
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06090539.html